CLINICAL TRIAL: NCT06079827
Title: Impact of Therapeutic Plasma Exchange on RNA Biomarker Expression Levels in Alzheimer's Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MaxWell Clinic, PLC (Industry)
Responsible Party: Sponsor
Other Study IDs: FBB-PE-003
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimens will be biobanked for potential follow up studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will determine if Therapeutic Plasma Exchange removes RNA biomarkers associated with Alzheimer's Disease and how quickly those biomarkers reappear after treatment.

DETAILED DESCRIPTION:
Participants with a diagnosis of Alzheimer's or Mild Cognitive Impairment will undergo therapeutic plasma exchange as part of their treatment for the disease as per the AMBAR Trial protocol. Patients will undergo one non-invasive tests to assess their microvascular system and complete one online test to assess the degree of cognitive impairment. Patients will have their blood drawn pre-plasma exchange, immediately post plasma exchange and repeated assessments and blood draws at seven day intervals post plasma exchange ending on the twenty-eighth day after the plasma exchange.

Their blood will be analyzed by FBB Biomed to identify the presence of unique RNA biomarkers associated with Alzheimer's disease and determine how quickly they regenerate.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is scheduled to undergo their first TPE Procedure for a diagnosis of Alzheimer's Disease or previous mental/cognitive impairment
2. Mentally capable of understanding and completing informed consent for the study.

Exclusion Criteria:

1. Subject is unable or failed to return/provide blood specimen on days seven (7), fourteen (14) , twenty-one (21), and twenty-eight (28) (plus or minus 1 day on follow up draws) post plasma exchange
2. Subject is unable to provide informed consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult individuals diagnosed with Alzheimer's Disease or mild cognitive impairment who will be undergoing plasma exchange per the AMBAR Trial protocol
Sampling Method: Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
To ascertain if Therapeutic Plasma Exchange (TPE) reduces the presence of RNA biomarkers in a small sample of Alzheimer's patients. | 28 days
  Measurement of RNA Biomarkers inside the participants blood stream

CONTACTS AND LOCATIONS:
Locations (1):
- The MaxWell Clinic, Brentwood, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Study results will be shared via publication to peer reviewed journals on Alzheimer's Disease and Cellular Medicine
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2-3 Years of study completion. Enduring in journal publication.